CLINICAL TRIAL: NCT06584136
Title: Lagged Relationships Between Sleep, Balance, and Cognition in Older Adults
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202302147
Record Dates: First submitted 2024-08-14; First posted 2024-09-04 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2024-12

CONDITIONS: Aging
Keywords: Sleep Quality; Balance Assessment; Older Adults; Cognitive Function; Sleep Monitoring; Wearable device
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oura ring: All participants will be assigned to a single group receiving a smart ring paired with their phone monitoring sleep and daily activity.

SUMMARY:
This study investigates the use of wearable devices and a sleep diary for tracking sleep and its impact on cognition and balance in older adults over six weeks. It will include routine mobility, balance assessment, and cognitive evaluations, focusing on analyzing the relationships between sleep, mobility, balance, and cognition.

DETAILED DESCRIPTION:
The study is designed to assess the relationships between sleep quality, balance capabilities, and cognitive functions in older adults. Using a longitudinal approach, participants will be monitored over six weeks with the help of wearable technology (OURA ring) and standardized assessments. Weekly in-person visits will include balance assessments using the Mini-BESTest and mobility tests such as the Timed Up and Go (TUG) test. Cognitive functions will be evaluated using the NIH Toolbox Cognitive Battery. The study aims to identify key sleep indicators that influence balance and cognition, ultimately contributing to improved strategies for maintaining the health and well-being of older adults.

ELIGIBILITY:
Inclusion Criteria:

Healthy older adults aged 65 and above English-speaking Independent in daily activities Able to walk independently or with minimal assistance (cane or walker) Willing to perform weekly assessments in balance and cognition at the University of Florida, Technology for Occupational Performance Lab

Exclusion Criteria:

Severe cognitive impairment (e.g., diagnosed dementia) Severe sleep disorders (e.g., sleep apnea requiring CPAP) Significant neurological conditions (e.g., Parkinson disease, stroke) Unstable medical conditions (e.g., uncontrolled hypertension, recent surgeries)

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy older adults aged 65 and above were recruited from the University of Florida, local retirement communities, and other relevant sources. They were without severe sleep disorders, cognitive impairment, Significant neurological conditions, or balance impairment.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time | 6-week daily assessments
  Total Sleep Time will be monitored using the OURA ring, calculated as the sum of all sleep stages in minutes each night. Data will be aggregated to provide a daily and weekly average for each participant.
Sleep Onset Latency | Daily assessments over 6 weeks
  Sleep Onset Latency, defined as the time taken to transition from wakefulness to sleep, will be recorded by the OURA ring each night. Data will be shown in daily and weekly for each participant.
Sleep Efficiency | Daily assessments over 6 weeks
  Sleep Efficiency will be measured as the ratio of total sleep time to time in bed, expressed as a percentage. The OURA ring will track this nightly, and the data will be summarized as daily data points and a weekly average.
Cognitive Function | 6 weeks weekly assessments
  Evaluated using the NIH Toolbox Cognitive Battery, with attention to memory, attention, and processing speed.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) Score | Pre-intervention (Baseline) and Post-intervention (Week 6)
  The Berg Balance Scale (BBS) will be administered twice, at baseline and at the end of the study period (Week 6), to assess changes in balance performance. The Berg Balance Scale (or BBS) is a widely used clinical test of a person&amp;amp;amp;amp;#39;s static and dynamic balance abilities.
Mini-BESTest Score | Weekly assessments over 6 weeks
  The Mini-BESTest will be conducted weekly throughout the 6-week study period to evaluate changes in balance performance over time. This test measures dynamic balance, functional mobility, and gait.
Daily Step Count | Daily assessments over 6 weeks recorded by Oura ring
  Daily step count will be monitored using the OURA ring. The data will be aggregated daily and weekly for each participant to assess overall physical activity levels.
Toe Strength from ToeScale | 6 weeks weekly assessments
  Measured using the ToeScale for both flexion and extension strength, comparing baseline and post-intervention data.

OTHER OUTCOMES:
Demographic Variables | Week 1 one time measured
  Demographic data, including age, gender, pre-existing conditions, and medical history, will be collected at the baseline (before the intervention begins). This data will be used to analyze participant characteristics and potential correlations with outcome measures.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data might be shared with permission from the funder and PI per request.
Supporting Information: Study Protocol
Time Frame: After study completion and publication of primary outcomes.
Access Criteria: Only de-identified data will be shared with permission from the funder and PI per request.
URL: https://top.ot.phhp.ufl.edu